CLINICAL TRIAL: NCT06280417
Title: Unreamed Intramedullary Tibial Nailing in Treatment of Open IIIa Diaphyseal Tibial Fractures in Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Ramzy Roshdy, Dr, Assiut University
Other Study IDs: Unreamed IMN In IIIa tibia
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Tibia Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Unreamed intramedullary tibial nail — Fixation of type IIIa tibial fractures by unreamed IMN

SUMMARY:
To study the incidence of non union of Unreamed intramedullary nailing in type IIIa Open diaphyseal fractures of the tibia as a primary outcome and the incidence of complications and clinical and functional outcome as a secondary outcome .

DETAILED DESCRIPTION:
Tibia is one of the most common bones to sustain open injury because of its superficial nature.Concerns over the high rates of malunion, nonunion, and deep infection have resulted in the development of aggressive treatment protocols including emergent wound exploration, thorough irrigation and debridement, bony stabilization, judicious antibiotic therapy, repeated wound debridements, and early soft-tissue coverage. However, there is still controversy regarding the optimal method of skeletal stabilization. High rates of pin tract infections, poor patient compliance, and malunion rates of 20% and greater have limited the use of external fixators as a definitive form of fixation.Despite initial encouraging results, plate fixation of open tibial fractures has been associated with implant failures, nonunions, and deep infection rates as high as 35%.6As a result, locked intramedullary nailing has become the standard treatment for open tibia fractures enabling axial alignment, early weight bearing, and immediate knee and ankle motion. Despite this, the complications including a high incidence of local bony necrosis and sepsis that occur following reamed intramedullary nails have led some to discourage the use of this method of skeletal stabilization in open tibia fractures.intramedullary tibial nail insertion without reaming has the advantage of minimal endosteal blood supply disruption and thus supposed to have increased union rate and reduction of infection rate .

Sanders et al 11 reported on the treatment of 64 patients with open tibial shaft fractures using unreamed interlocked intramedullary nails. All but 1 of the fractures healed with excellent alignment and an overall chronic infection rate of 4%.other studies reported similar results .12 type and timing of fixation were important determinants of infection , with people who received intramedullary nailing within 24 h having the lowest risk of infection .UTN significantly reduced the incidence rates of superficial infection and malunion compared with EF, suggesting that it is likely a safe and effective alternative to EF for treating open tibial fractures. however patients' postoperative weight bearing should be controlled to avoid hardware failure.

Here,our purpose is to investigate the outcome of Unreamed intramedullary nail in open diaphyseal fractures of the tibia in our setup .

ELIGIBILITY:
Inclusion Criteria:

1. Open grade IIIa diaphyseal tibial fractures .
2. Skeletaly mature patients .

Exclusion Criteria:

1. late presentation and open infected fractures .
2. Associated intraarticular fractures of proximal /distal tibia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with type IIIa diaphyseal tibial fractures are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of non union | Baseline
  Preoperative and postoperative x-ray anteroposterior & lateral views including both ankle and knee joints

SECONDARY OUTCOMES:
Incidince of fracture related infection | Baseline
  Culture and sensitivity and blood tests
The rate of reoperation for delayed union or non-union , infection and fasciotomy | Baseline
functional evaluation | Baseline
  Modified Karlstrom- Olerud Score

REFERENCES:
- [Background] Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial Fractures Investigators; Bhandari M, Guyatt G, Tornetta P 3rd, Schemitsch EH, Swiontkowski M, Sanders D, Walter SD. Randomized trial of reamed and unreamed intramedullary nailing of tibial shaft fractures. J Bone Joint Surg Am. 2008 Dec;90(12):2567-78. doi: 10.2106/JBJS.G.01694. PMID 19047701
- [Background] Rhinelander FW. Tibial blood supply in relation to fracture healing. Clin Orthop Relat Res. 1974 Nov-Dec;(105):34-81. No abstract available. PMID 4609655
- [Background] Henley MB, Chapman JR, Agel J, Harvey EJ, Whorton AM, Swiontkowski MF. Treatment of type II, IIIA, and IIIB open fractures of the tibial shaft: a prospective comparison of unreamed interlocking intramedullary nails and half-pin external fixators. J Orthop Trauma. 1998 Jan;12(1):1-7. doi: 10.1097/00005131-199801000-00001. PMID 9447512
- [Background] Edwards CC, Simmons SC, Browner BD, Weigel MC. Severe open tibial fractures. Results treating 202 injuries with external fixation. Clin Orthop Relat Res. 1988 May;(230):98-115. PMID 3365903
- [Background] Bach AW, Hansen ST Jr. Plates versus external fixation in severe open tibial shaft fractures. A randomized trial. Clin Orthop Relat Res. 1989 Apr;(241):89-94. PMID 2924483
- [Background] Bone LB, Johnson KD. Treatment of tibial fractures by reaming and intramedullary nailing. J Bone Joint Surg Am. 1986 Jul;68(6):877-87. PMID 3733776
- [Background] Larsen LB, Madsen JE, Hoiness PR, Ovre S. Should insertion of intramedullary nails for tibial fractures be with or without reaming? A prospective, randomized study with 3.8 years' follow-up. J Orthop Trauma. 2004 Mar;18(3):144-9. doi: 10.1097/00005131-200403000-00003. PMID 15091267
- [Background] Gustilo RB, Mendoza RM, Williams DN. Problems in the management of type III (severe) open fractures: a new classification of type III open fractures. J Trauma. 1984 Aug;24(8):742-6. doi: 10.1097/00005373-198408000-00009. PMID 6471139
- [Background] Sanders R, Jersinovich I, Anglen J, DiPasquale T, Herscovici D Jr. The treatment of open tibial shaft fractures using an interlocked intramedullary nail without reaming. J Orthop Trauma. 1994 Dec;8(6):504-10. PMID 7869165
- [Background] Joshi D, Ahmed A, Krishna L, Lal Y. Unreamed interlocking nailing in open fractures of tibia. J Orthop Surg (Hong Kong). 2004 Dec;12(2):216-21. doi: 10.1177/230949900401200215. PMID 15621910
- [Background] Schade AT, Sabawo M, Nyamulani N, Mpanga CC, Ngoie LB, Metcalfe AJ, Lalloo DG, Madan JJ, Harrison WJ, MacPherson P. Functional outcomes and quality of life at 1-year follow-up after an open tibia fracture in Malawi: a multicentre, prospective cohort study. Lancet Glob Health. 2023 Oct;11(10):e1609-e1618. doi: 10.1016/S2214-109X(23)00346-7. Epub 2023 Sep 1. PMID 37666261
- [Background] Fu Q, Zhu L, Lu J, Ma J, Chen A. External Fixation versus Unreamed Tibial Intramedullary Nailing for Open Tibial Fractures: A Meta-analysis of Randomized Controlled Trials. Sci Rep. 2018 Aug 24;8(1):12753. doi: 10.1038/s41598-018-30716-y. PMID 30143702
- [Background] Mohseni MA, Soleimanpour J, Mohammadpour H, Shahsavari A. AO tubular external fixation vs. unreamed intramedullary nailing in open grade IIIA-IIIB tibial shaft fractures: a single-center randomized clinical trial. Pak J Biol Sci. 2011 Apr 15;14(8):490-5. doi: 10.3923/pjbs.2011.490.495. PMID 21936253